CLINICAL TRIAL: NCT04417686
Title: ARTERIAL EMBOLIZATION OF PERSISTENT GENICULATE ARTERIES FOR CHRONIC PAIN MANAGEMENT AFTER TOTAL KNEE-REPLACEMENT ARTHROPLASTY: A FEASIBILITY STUDY (KNEE EMBOLISATION)
Brief Title: ARTERIAL EMBOLIZATION OF PERSISTENT GENICULATE ARTERIES FOR CHRONIC PAIN MANAGEMENT AFTER TOTAL KNEE-REPLACEMENT ARTHROPLASTY(KNEE EMBOLISATION)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-22; 2019-A00746-51 (Other: IDRCB)
Record Dates: First submitted 2020-06-02; First posted 2020-06-05 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Musculoskeletal Inflammatory

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patient (Experimental)
  Interventions: Procedure: arterial embolization

INTERVENTIONS:
Procedure: arterial embolization — arterial embolization of the geniculated arteries for reduction of pain after installation of total knee prosthesis

SUMMARY:
Recent works in interventional radiology have shown interesting results in the treatment of musculoskeletal inflammatory sites by arterial embolization. Supra-selective arterial embolization has been successfully developed by Dr. Okuno (Japan) to manage moderate to severe knee osteoarthritis. Also, inflammation of the surgical site mediated via geniculate arteries is a major cause for persistent chronic post-operative gonalgia.

DETAILED DESCRIPTION:
Hypothesis: Selective arterial embolization of persistent geniculate arteries could reduce chronic post-operative gonalgia after TKA with minimally invasive approach.

Objective: To evaluate the feasibility of selective arterial embolization of persistent geniculate arteries to reduce chronic post-operative gonalgia after TKA.

Material and methods: This study is a single-center, prospective, feasibility study. Patients will be recruited after rheumatology consultation for chronic post-operative gonalgia, more than 6 months after TKA for moderate to severe gonarthrosis. Eligible patients are adults with moderate to severe chronic post-operative gonalgia (Visual Analysis Scale (VAS) > 50mm) and degraded life quality (assessed by SF36 score), despite at least 3 months of optimal medical treatment. Non-inclusion criteria are mainly other rheumatologic or orthopedic severe diseases, severe surgical complications. Under local anesthesia, with homolateral antegrade femoral access, patient will undergo selective arterial embolization of persistent and aberrant peri-prosthetic arteries using HydroPearl® 200µm Mircospheres. Follow-up consultations will be scheduled at D1, M1, M3, M6 and M12. For a significance level of α=0.05 and power of 80% we require a cohort of 24 patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (male or female) aged 18-85
* Suffering from moderate to severe chronic pain (EVA > 50mm) more than 6 months after total prosthetic knee replacement surgery for severe gonarthrosis with impact on quality of life.
* And having followed for at least 3 months a well-conducted conservative medical treatment (anti-inflammatory, analgesic, masso-kinesiotherapy).
* The patient may initially have had a single or bilateral replacement. The period of 6 months must be respected for each side, between the intervention and the inclusion for homolateral pain.
* Patient willing to participate in the study and with signed informed consent.
* Patient willing to undergo post-operative monitoring for one year.

Exclusion Criteria:

Orthopaedic or rheumatological pathologies:

* Rheumatoid arthritis
* Psoriatic rheumatism
* Spondylarthropathies
* History of primary or secondary bone tumor, in remission or active.
* Myeloma
* Operational criteria:
* Infection of the surgical site
* Re-operation
* Severe bleeding
* Use of turnstile per-operative
* Wound of popliteal artery
* Diabetic patient
* Comorbidities:
* General condition responsible for objective hemostasis disorder (hemophilia, Willebrand disease, thrombocytopenia) and anticoagulant treatments.
* Pads 100 G/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-06-22 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
arterial embolization | 12 MONTHS

SECONDARY OUTCOMES:
VAS pain score | 12MONTHS
Western Ontario and Universities Osteroarthritis Index (WOMAC) score | 12MONTHS
SF36 quality of life score | 12 MONTHS

CONTACTS AND LOCATIONS:
Overall Officials: EMILIE GARRIDO PRADALIE, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France